CLINICAL TRIAL: NCT06142344
Title: The Added Value of 166Ho Trans-arterial Radioembolization to Systemic Therapy in Liver Metastatic Breast Cancer Patients
Brief Title: Radioembolisation and Chemotherapy in Liver Metastatic Breast Cancer Patients
Acronym: HoLiBreast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21RTA
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Liver Metastases; Breast Cancer
Keywords: Liver metastatic breast cancer; Holmium-166; Radioembolization; TARE; SIRT; Selective internal radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ho-166 radioembolization (Experimental): Patients will undergo standard procedures for holmium radioembolization
  Interventions: Device: Quiremspheres™

INTERVENTIONS:
Device: Quiremspheres™ — The intervention comprises two steps. Initially, the patient will undergo mapping angiography and a Ho-166 scout dose. If deemed eligible, the patient will proceed to 166-Ho radioembolization.
  Other Names: Radioembolization with Quiremspheres™

SUMMARY:
The goal of this multicentre clinical pilot study is to investigate the feasibility of the addition of Ho-166 radioembolization to chemotherapy in patients with liver metastastic breast cancer.

Participants will receive a mapping angiography and Ho-166 radioembolization. Chemotherapy will be stopped 2-5 prior to radioembolization and continuation of chemotherapy will be evaluated at 2 weeks post-radioembolization.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years
* Patients with hormone positive and HER2 negative liver metastatic breast cancer
* No extra-hepatic disease progression at evaluation of at least second line systemic chemotherapy
* Suitable for TARE evaluated after the mapping angiography
* Measurable target tumors in the liver according to RECIST 1.1
* Liver tumor burden <50 %
* ECOG performance score 0 to 1
* Laboratory parameters: neutrophils >1000/μL; thrombocyte count >1000000 μL; eGFR >45/mL/min/1.73 m2; albumin > 3.0 g/dl, bilirubin < 1.5x ULN (unless Gilbert syndrome); aminotransferase (ALAT/ASAT) <3.0 ULN
* Able to read Dutch

Exclusion Criteria:

* Life expectancy ≤3 months
* Patient eligible for other curative local liver therapy (ea. surgery, ablation)
* Brain, pleural, peritoneal or extensive extra-hepatic visceral metastases
* Other life-threatening disease (i.e. Dialysis, unresolved diarrhea, serious unresolved infections (HIV, HBV, HCV etc.))
* Contraindication for angiography or MRI
* Significant toxicities due to prior cancer therapy that have not resolved before the initiation of the study, if the investigator determines that the continuing complication will compromise the safe treatment of the patient
* Prior or planned embolic intra-arterial liver directed therapy (TACE, TAE, TARE)
* Prior or planned external or internal radiation therapy of the liver
* Cirrhosis or portal hypertension
* Main portal vein thrombosis
* Intervention for, or compromise of, the Ampulla of Vater
* Ascites (except minor focal ascites)
* Baseline use of analgesics for abdominal pain
* Pregnancy (Women at childbearing potential need at least one form of birth control) and breastfeeding
* Flow to extra hepatic vessels not correctable by reposition or embolization
* Estimated dose to the lungs greater than 30 Gy in a single administration or 50 Gy cumulatively
* Target tumoral absorbed dose of < 90Gy or an absorbed dose to the normal liver parenchyma of >50Gy (in case of whole liver treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Up to 3 months after intervention
  The percentage of patients were radioembolization and systemic chemotherapy is safely feasible. Safety is defined as percentage of 90 day post-radioembolization (CTCAE/SIR grade 3 or higher) which lead discontinuation of the current systemic chemotherapy. Time to re-start chemotherapy after intervention in days will be collected.

SECONDARY OUTCOMES:
Lesion- and patient-based response | Up to 3 months after intervention
  Radiological response on contrast-enhanced CT and MRI measured by RECIST
Overall toxicity associated with study intervention | Up to 3 months after intervention
  Graded by CTCAE/SIR grade
Quality of Life during study | From start inclusion to 3 months after intervention
  Obtained by EORTC QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No